CLINICAL TRIAL: NCT00967525
Title: A Pilot Study of Intraosseous Infusion of Unrelated Cord Blood Grafts
Brief Title: Intraosseous Infusion of Unrelated Cord Blood Grafts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Horan, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000113; Intraosseous Infusion (Other: Other)
Record Dates: First submitted 2009-08-11; First posted 2009-08-28 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; ALL; leukemia; CML; Myelodysplastic Syndrome; malignancies; Undifferentiated leukemia; High risk malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receive two cord blood units. One administered by intraosseous infusion and the other by intravenous infusion. The second unit is being given as a safeguard, but will also allow the researchers to directly compare engraftment between intravenously and intraosseously infused cord blood units.
  Interventions: Procedure: cord blood infusion

INTERVENTIONS:
Procedure: cord blood infusion — Receive two cord blood units. One administered by intraosseous infusion and the other by intravenous infusion. The second unit is being given as a safeguard, but will also allow the researchers to directly compare engraftment between intravenously and intraosseously infused cord blood units.

SUMMARY:
In this trial the investigators seek to determine if injecting cord blood cells directly into the bone marrow (intraosseous injection), rather than infusing them intravenously, can improve engraftment. The rational for doing this is that most hematopoietic stem cells (HSCs) infused intravenously never reach the bone marrow, getting trapped by other organs, such as the lungs, instead. The potential advantage of intraosseous infusion is suggested by studies in rodents that have demonstrated that in HSC transplants where the cell dose is limiting intraosseous injection is a more effective route of administration. The safety of intraosseous injections, in general, is underscored by the vast experience using intraosseous injections for resuscitation of critically ill children. The safety of injecting HSCs intraosseously has been demonstrated in a clinical trial of transplanting bone marrow cells.

To safeguard against problems that might result, if intraosseous infusion fails to improve engraftment in this trial, the investigators will integrate a recently introduced strategy proven to improve engraftment-the transplantation of two cord blood units. Transplanting two unrelated cord blood units by intravenous infusion has been shown to improve engraftment (although there is still room for improvement). In this trial one unit will be injected intraosseously and the other unit will be infused intravenously.

This study is being conducted as a forerunner to a larger, multi-center trial. The investigators intend to enroll five patients over 1-2 years.

DETAILED DESCRIPTION:
Hematopoietic (blood forming) stem cells (HSCs) reside primarily in the bone marrow. Traditionally, HSCs have been obtained directly from the bone marrow. Transplants using cells obtained this way are referred to as bone marrow transplants. HSCs also circulate in the blood. Transplants using cells obtained from the blood of children and adults are referred to as peripheral blood stem cell transplants. The blood of fetuses is especially rich in HSCs and these cells can be easily collected at birth from the placenta. Transplants using these cells are called cord blood transplants. Although HSCs can be collected from various sites, all HSC transplants, regardless of the source, are given to recipients by intravenous infusion. The transplanted HSCs then migrate to the bone marrow.

Over the past ten years unrelated cord blood transplantation has become an accepted alternative to bone marrow transplantation. African-Americans and other minorities, who are underrepresented in the National Marrow Donor Program, have benefited particularly from this. In infants and young children cord blood transplantation appears to be as effective as bone marrow transplantation. In older children, adolescents and adults, however, cord blood transplantation has not been as effective, primarily because most cord blood units provide an insufficient number of cells to ensure prompt and reliable engraftment ("taking" of the transplanted cells in the recipient's bone marrow).

ELIGIBILITY:
Inclusion Criteria:

1. Age 36 months to 60 years old (YO)
2. No prior autologous or allogeneic transplant
3. Karnofsky performance score or Lansky Play-Performance of at least 80

Exclusion Criteria:

1. Age < 36 months or > 60 YO
2. creatinine clearance or nuclear medicine GFR of < 50 mL/min
3. cardiac ejection fraction < 50%
4. bilirubin > 2 × upper limit of normal or ALT > 4 × upper limit of normal or unresolved veno-occlusive disease
5. Pulmonary carbon monoxide diffusing capacity (DLCO), adjusted for Hgb < 50%
6. Karnofsky performance score or Lansky Play-Performance Scale <80
7. Uncontrolled viral, bacterial, or fungal infection at the time of study enrollment
8. Seropositive for HIV
9. Availability of a willing and well HLA matched related (genotypically identical or mismatched at a single allele or antigen defined by typing at HLA A, B, C and DRB1 loci) donor
10. Availability of a willing and well HLA matched unrelated (allele matched or mismatched at a single allele defined by allele level typing for HLA A, B, C and DRB1 loci) adult blood or marrow donor
11. Availability of an umbilical cord blood unit, which provides at least a 4/6 HLA match as defined above and ≥ 5.0 * 107 NC/Kg (cryopreserved)

Ages: 36 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Compare the rapidity of myeloid engraftment of intraosseously and intravenously administered unrelated cord blood grafts. | 1 year after last patient enrolled

SECONDARY OUTCOMES:
Obtain preliminary data using flow cytometric analysis to assess the importance of graft associated variables that may affect engraftment. | 1 year after last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: John Horan, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia